CLINICAL TRIAL: NCT05681975
Title: Food-specific Immunoglobulin G4 and Immunoglobulin E Antibody Reactions in a Population With Adverse Reactions to Foodstuffs-related Symptoms
Brief Title: Immunoglobulin G4 and Immunoglobulin E Antibodies in a Population With Adverse Reactions to Foodstuffs-related Symptoms
Status: Recruiting | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Lisset Pantoja Arevalo, Food Engineer, Master of Food Engineering applied to health, Universidad Politecnica de Madrid
Other Study IDs: 1720IL0389
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Immunoglobulin E-Mediated Food Allergy; Immunoglobulin G4-Related Disease; Symptoms and Signs; Adverse Reaction to Food
MeSH Terms: conditions — Food Hypersensitivity; Immunoglobulin G4-Related Disease; Signs and Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Capillary whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Food-specific Immunoglobulin G4 and/or Immunoglobulin E antibody reactions — Immunoassay kits (NutriSMART® and Fastcheckpoc20® In-Vitro Diagnostic kits, DST GmbH, Schwerin, Germany) are performed in a population with suspicion of having a food allergy or a food intolerance with related symptoms.

SUMMARY:
The aim of this study is to analyze a population with symptoms associated with adverse reactions to foodstuffs (ARFS). To determine the levels of food-specific immunoglobulin G4 (IgG4) and immunoglobulin E (IgE) antibody reactions (AbR).

DETAILED DESCRIPTION:
Volunteers with symptoms related with adverse reactions to foodstuffs (ARFS) and suspicion of having a food allergy or a food intolerance are enrolled in this study. A 50μl of capillary whole blood is analyzed and the levels of food-specific immunoglobulin G4 (IgG4) or immunoglobulin E (IgE) antibody reactions (AbR) are determined.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* To present symptoms related to adverse reactions to foodstuffs (ARFS)

Exclusion Criteria:

* Antibiotic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults presenting symptoms related to adverse reactions to foodstuffs and/ or with suspicion of having a food allergy or food intolerance
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Food-specific Immunoglobulin G4 antibody reactions | 0 days
  Immunoassay kits (NutriSMART® In-Vitro Diagnostic kit, DST GmbH, Schwerin, Germany) are performed in a population with suspicion of having a food allergy or a food intolerance with related symptoms.

SECONDARY OUTCOMES:
Food-specific Immunoglobulin E antibody reactions | 0 days
  Immunoassay kits (Fastcheckpoc20® In-Vitro Diagnostic kit, DST GmbH, Schwerin, Germany) are performed in a population with suspicion of having a food allergy or a food intolerance with related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lisset Pantoja-Arévalo, MSc, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided